CLINICAL TRIAL: NCT02728570
Title: Effect of Dietary Flavonoids on Intestinal Microbiota, Intestinal Inflammation and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: USU #5483
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Metabolic Syndrome X; Inflammation
Keywords: flavonoids; insulin resistance; plasma lipids; intestinal microbiome; intestinal inflammation; subclinical inflammation
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Flavonoids then High Flavonoids (Experimental): Participants receive a prepared diet with Low Dietary Flavonoids (10 mg of flavonoids/1000 Kcals) for six weeks. After a minimum washout period of 2 weeks, participants receive a prepared diet with High Dietary Flavonoids (340 mg of flavonoids/1000 Kcals) for six weeks.
  Interventions: Other: High Dietary Flavonoids; Other: Low Dietary Flavonoids
- High Flavonoids then Low Flavonoids (Experimental): Participants receive a prepared diet with High Dietary Flavonoids (340 mg of flavonoids/1000 Kcals) for six weeks. After a minimum washout period of 2 weeks, participants receive a prepared diet with Low Dietary Flavonoids (10 mg of flavonoids/1000 Kcals) for six weeks.
  Interventions: Other: High Dietary Flavonoids; Other: Low Dietary Flavonoids

INTERVENTIONS:
Other: High Dietary Flavonoids — A prepared diet consisting of whole foods with a macronutrient composition of 17% en from protein, 30% en from fat and 53% energy from carbohydrate and containing high levels of dietary flavonoids including anthocyanins, flavanones, flavan-3-ols, flavonols, flavones, and polyflavonoids.
Other: Low Dietary Flavonoids — A prepared diet consisting of whole foods with a macronutrient composition of 17% en from protein, 30% en from fat and 53% energy from carbohydrate and containing low levels of dietary flavonoids including anthocyanins, flavanones, flavan-3-ols, flavonols, flavones, and polyflavonoids.

SUMMARY:
The investigators have hypothesized that dietary flavonoids reduce insulin resistance and subclinical inflammation secondary to reductions in intestinal inflammation and permeability and that these events are mediated through alterations in gut microbiota composition. To test this hypothesis, 30 overweight/obese men and women will be provided two well-controlled diets that are identical in macronutrient content (Protein, 17% en; Fat, 30% en; Carbohydrate, 53% en), but differ markedly in flavonoid content (Low Flavonoid Diet, 10 mg/1000 Kcals; High Flavonoid Diet, 340 mg/1000 Kcals). All meals for both diets will be prepared and fed for 6 weeks each in a randomized cross-over design with endpoints determined in duplicate during the last week of each diet period.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kg/m2

Exclusion Criteria:

* Documented presence of atherosclerotic disease;
* Diabetes mellitus
* Uncontrolled hypertension
* Renal, hepatic, endocrine, gastrointestinal or other systemic disease
* For women, pregnancy, breast feeding or postpartum < 6 months
* History of drug or alcohol abuse
* History of depression or mental illness requiring hospitalization within the last 12 months
* Use of antibiotics within the last 6 months
* Multiple food allergies or significant food preferences or restrictions that would interfere with diet adherence
* Chronic use of over-the-counter medication which would interfere with study endpoints including NSAIDS, laxatives and antacids
* Lifestyle or schedule incompatible with the study protocol
* Other medical, psychiatric, or behavioral conditions that in the view of the principal investigator may present a safety hazard to the participant or interfere with study participation or the ability to follow the intervention protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Fecal calprotectin | 6 weeks
  Primary endpoint for intestinal inflammation
Serum C-reactive protein | 6 weeks
  One of two primary endpoints for systemic inflammation
Serum soluble tumor necrosis factor receptor-1 | 6 weeks
  One of two primary endpoints for systemic inflammation
Serum insulin | 6 weeks
  Primary endpoint for insulin resistance

SECONDARY OUTCOMES:
Fecal microbiome composition | 6 weeks
  Includes relative abundances of operational taxonomic units and assigned taxonomy as well as alpha and beta diversity measurements
Fecal short chain fatty acids | 6 weeks
  Measure of fecal microbiome metabolic capabilities and includes acetate, propionate, butyrate, valerate and caproate.
Fecal eosinophil protein X | 6 weeks
  Secondary endpoint for intestinal inflammation
Fecal myeloperoxidase | 6 weeks
  Secondary endpoint for intestinal inflammation
Intestinal permeability by four sugar differential absorption test | 6 weeks
  Secondary endpoint for intestinal inflammation
Serum endotoxin | 6 weeks
  Secondary endpoint for intestinal inflammation
Serum interleukin-6 | 6 weeks
  Secondary endpoint for systemic inflammation
Serum soluble tumor necrosis factor receptor-2 | 6 weeks
  Secondary endpoint for systemic inflammation
Serum fasting glucose | 6 weeks
  Secondary endpoint for insulin resistance
Calculated Homeostatic Model Assessment-Insulin Resistance | 6 weeks
  Secondary endpoint for insulin resistance
Serum C-peptide | 6 weeks
  Secondary endpoint for insulin resistance
Plasma lipids | 6 weeks
  Secondary endpoint for insulin resistance. Includes LDL-cholesterol, HDL-cholesterol and triglycerides
Blood pressure | 6 weeks
  Secondary endpoint for insulin resistance. Includes systolic and diastolic blood pressure

OTHER OUTCOMES:
Serum resistin | 6 weeks
  Measure of adipocyte inflammation and systemic metabolism
Serum visfatin | 6 weeks
  Measure of adipocyte inflammation and systemic metabolism
Serum adiponectin | 6 weeks
  Measure of adipocyte inflammation and systemic metabolism
Serum leptin | 6 weeks
  Measure of adipocyte inflammation and systemic metabolism
Body weight | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lefevre, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be deposited into a public repository as the data are published.